CLINICAL TRIAL: NCT02040844
Title: An Optional Prospective Follow-on Study to Evaluate the Continued Efficacy and Safety of Cat-PAD in Cat Allergic Subjects up to Five Years After the Administration of Treatment
Brief Title: Phase III Cat-PAD Follow-on Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Circassia Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP007 A
Record Dates: First submitted 2014-01-17; First posted 2014-01-20 (Estimated); Results first posted 2018-05-14 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-05

CONDITIONS: Cat Allergy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cat-PAD Treatment 1 (Other): Received Cat-PAD Treatment 1 in Study CP007 [NCT01620762].No further treatment received in CP007A
  Interventions: Drug: Received Cat-PAD Treatment 1 in Study CP007 [NCT01620762]
- Cat-PAD Treatment 2 (Other): Received Cat-PAD Treatment 2 in Study CP007 [NCT01620762].No further treatment received in CP007A.
  Interventions: Drug: Received Cat-PAD Treatment 2 in Study CP007 [NCT01620762]
- Cat-PAD Treatment 3 (Other): Received Cat-PAD Treatment 3 in Study CP007 [NCT01620762]. No further treatment received in CP007A.
  Interventions: Drug: Received Cat-PAD Treatment 3 in Study CP007 [NCT01620762]

INTERVENTIONS:
Drug: Received Cat-PAD Treatment 1 in Study CP007 [NCT01620762]
  Arms: Cat-PAD Treatment 1
Drug: Received Cat-PAD Treatment 2 in Study CP007 [NCT01620762]
  Arms: Cat-PAD Treatment 2
Drug: Received Cat-PAD Treatment 3 in Study CP007 [NCT01620762]
  Arms: Cat-PAD Treatment 3

SUMMARY:
The purpose of this study is to evaluate the continued effectiveness and safety of Cat-PAD in cat allergic subjects for up to five years after the start of administration of treatment. The study is an optional follow-up study to a phase III double-blind, placebo controlled, Cat-PAD study; no further investigational product is administered.

ELIGIBILITY:
Inclusion Criteria:

* previously completed clinical study CP007 [NCT01620762]

Exclusion Criteria:

* started allergen therapy since completing CP007
* Institutionalised due to a legal or regulatory order

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Kleine-Tebbe, MD, Principal Investigator — Clinical Research Center for Dermatology, Allergy & Asthma

RESULTS

PARTICIPANT FLOW:
Groups:
- Cat-PAD Treatment 1 (1 Course): Cat-PAD: 1 dose every 4 weeks followed by placebo 1 dose every 4 weeks
- Cat-PAD Treatment (2 Courses): Cat-PAD: 1 dose every 4 weeks followed by a second course of 1 dose every 4 weeks
- Placebo: Placebo - 1 dose every 4 weeks
Period: Overall Study
Arm/Group | Cat-PAD Treatment 1 (1 Course) | Cat-PAD Treatment (2 Courses) | Placebo
Started | 138 | 148 | 144
Completed | 88 | 109 | 97
Not Completed | 50 | 39 | 47
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Withdrawal by Subject | 16 | 22 | 25
Not completed — Lost to Follow-up | 12 | 9 | 13
Not completed — Missing | 13 | 3 | 2
Not completed — Non-specified | 8 | 2 | 5
Not completed — Concomitant medication | 1 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cat-PAD Treatment 1 (1 Course) | Cat-PAD Treatment (2 Courses) | Placebo | Total
Number analyzed (Participants) | 138 | 148 | 144 | 430
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 10 | 8 | 23
  Between 18 and 65 years | 133 | 137 | 135 | 405
  >=65 years | 0 | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 106 | 97 | 292
  Male | 49 | 42 | 47 | 138
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 135 | 145 | 139 | 419
  Black | 2 | 1 | 1 | 4
  Asian (Indian) | 0 | 1 | 0 | 1
  Asian (Oriental) | 0 | 0 | 3 | 3
  American hispanic | 0 | 1 | 1 | 2
  Other | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: Subjects]
  United States | 31 | 30 | 41 | 102
  Europe | 68 | 82 | 68 | 218
  Canada | 39 | 36 | 35 | 110

OUTCOME MEASURES:

1. Primary Outcome: Mean Combined Score (CS) Consisting of TRSS/8+Allergy Medication Score[AMS])
Description: The primary endpoint was the mean Combined Score (CS) in Cat-PAD treatment groups compared with the mean CS in the placebo group. This was assessed one year after completing the original study (CP007).
  CS = Total Rhinoconjunctivitis Symptom Score (TRSS) + Allergy Medication Score (AMS). Eight symptoms are defined in the TRSS, 4 nasal symptoms: runny nose, sneezing; blocked nose and itchy nose and 4 ocular symptoms: itchy eyes; watery eyes; red eyes and sore eyes. Each symptom was rated in severity on a score of 0-3 (0=absent, 3=severe) and the TRSS was divided by the number of symptoms to provide an average score per symptom of 0-3.
  AMS was scored from 0 (no allergy rescue medication use per day) to 3 (at least one dose of systemic corticosteroid per day). The AMS score was not additive, and therefore the maximum AMS was 3 and the maximum CS was 6.
Time Frame: 1 year after completing CP007
Population: The number of subjects included in the analysis is the total number of subjects that completed the End of Year 1 assessments (1 year after the completion of CP007 and 2 years after the start of treatment).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Cat-PAD Treatment 1 (1 Course) | Cat-PAD Treatment (2 Courses) | Placebo
Number analyzed (Participants) | 88 | 109 | 97
units on a scale | 1.99 (0.16) | 1.91 (0.15) | 1.93 (0.15)

2. Secondary Outcome: Mean TRSS
Description: Mean Total Rhinoconjunctivitis Symptom Score (TRSS) in Cat-PAD treatment groups compared with placebo.
  Eight symptoms are defined in the TRSS, 4 nasal symptoms: runny nose, sneezing; blocked nose, and itchy nose and 4 ocular symptoms: itchy eyes; watery eyes; red eyes, and sore eyes. Each symptom was rated in severity on a score of 0-3 (0. absent; 1. mild, barely noticeable; 2. moderate, annoying/troublesome; 3. severe, very annoying/very troublesome), therefore TRSS could range from 0 to 24. Higher TRSS reflected more severe symptom scores. Symptoms were scored daily for a period of approximately 3 weeks one year after completing the first study (CP007).
Time Frame: 1 year after completion of CP007
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Cat-PAD Treatment 1 (1 Course) | Cat-PAD Treatment (2 Courses) | Placebo
Number analyzed (Participants) | 88 | 109 | 97
units on a scale | 12.95 (0.69) | 13.15 (0.66) | 12.92 (0.67)

3. Secondary Outcome: Mean Component Scores of the TRSS (Nasal)
Description: TNSS (Total nasal symptom score) was the sum of all the nasal symptom scores (runny nose; sneezing; blocked nose; itchy nose) and could range from 0 to 12. Higher TNSS reflected more severe symptoms.
  Subjects rated the severity of each symptom over the last 24 hours as follows: 0. absent; 1. mild, barely noticeable; 2. moderate, annoying/troublesome; 3. severe, very annoying/very troublesome. Symptoms were scored daily for a period of approximately 3 weeks 1 year after completing the original CP007 study.
Time Frame: 1 year after completion of CP007
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Cat-PAD Treatment 1 (1 Course) | Cat-PAD Treatment (2 Courses) | Placebo
Number analyzed (Participants) | 88 | 109 | 97
units on a scale | 7.06 (0.39) | 7.17 (0.37) | 6.96 (0.38)

4. Secondary Outcome: Mean Component Scores of the TRSS (Ocular)
Description: Mean daily Total Ocular Symptom Score (TOSS) in Cat-PAD treatment groups compared to placebo groups
  Eight symptoms are defined in the TRSS, 4 nasal symptoms: runny nose, sneezing; blocked nose, and itchy nose and 4 ocular symptoms: itchy eyes; watery eyes; red eyes, and sore eyes. TOSS was the sum of all the ocular symptom scores (itchy eyes; watery eyes; red eyes; sore eyes) and could range from 0 to 12. Higher TOSS reflected more severe symptoms.
  Subjects rated the severity of each symptom over the last 24 hours as follows: 0. absent; 1. mild, barely noticeable; 2. moderate, annoying/troublesome; 3. severe, very annoying/very troublesome. Symptoms were scored daily for a period of approximately 3 weeks one year after completing the original CP007 study
Time Frame: 1 year after completion of CP007
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Cat-PAD Treatment 1 (1 Course) | Cat-PAD Treatment (2 Courses) | Placebo
Number analyzed (Participants) | 88 | 109 | 97
units on a scale | 5.90 (0.35) | 5.97 (0.33) | 6.00 (0.34)

5. Secondary Outcome: Mean Allergy Medication Score (AMS)
Description: Mean AMS (Allergy medication score) in Cat-PAD treatment groups compared with placebo groups.
  The use of rhinoconjunctivitis rescue medications was recorded by the subject for a period of 21 days, on a daily basis just before bedtime, approximately 1 year after completing the original CP007 study. Rescue medication use was scored based on a previously published system as follows: 0 = no allergy rescue medication used per day; 0.5 = at least one dose of antihistamine eye drops used per day; 1 = at least one dose of oral antihistamine used per day; 2 = at least one dose of intranasal corticosteroid used per day; 3 = at least one dose of systemic corticosteroid used per day. The score was according to the highest level of rescue medication used and was not additive.
Time Frame: 1 year after completion of CP007
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Cat-PAD Treatment 1 (1 Course) | Cat-PAD Treatment (2 Courses) | Placebo
Number analyzed (Participants) | 88 | 109 | 97
units on a scale | 0.37 (0.09) | 0.27 (0.09) | 0.31 (0.09)

6. Secondary Outcome: Mean RQLQ Score
Description: The RQLQ (Rhinoconjunctivitis Quality of Life Questionnaire) was completed by subjects one year after the completion of the previous study (CP007).
  The RQLQ is a validated method of assessing quality of life and has 28 questions in seven domains (activity limitation, sleep problems, nasal symptoms, eye symptoms, non-nasal/eye symptoms, practical problems and emotional function). Subjects recalled how their rhinoconjunctivitis had been during the last week and responded to each question on a seven-point scale (0 = no impairment, 6 = maximum impairment). The questions were equally weighted, and the RQLQ score was the mean of the 28 questions and could range from zero to six.
  A higher score indicated greater impact on quality of life and thus a low score indicated a better outcome.
Time Frame: 1 year after completion of CP007
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Cat-PAD Treatment 1 (1 Course) | Cat-PAD Treatment (2 Courses) | Placebo
Number analyzed (Participants) | 88 | 109 | 97
units on a scale | 1.58 (0.22) | 1.62 (0.21) | 1.51 (0.22)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected throughout the whole study period from the point of enrolment to the completion of outcome data which was timed to occur 2 year after the completion of the original CP007 study
Arm/Group | Cat-PAD Treatment 1 (1 Course) | Cat-PAD Treatment (2 Courses) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/138 | 0/148 | 0/144
Serious Adverse Events (participants affected / at risk) | 3/138 | 4/148 | 3/144
Other Adverse Events (participants affected / at risk) | 54/138 | 62/148 | 56/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cat-PAD Treatment 1 (1 Course) (N=138) | Cat-PAD Treatment (2 Courses) (N=148) | Placebo (N=144)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Anapylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Colonic fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Colonic abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastronteritis Escheria coli (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cat-PAD Treatment 1 (1 Course) (N=138) | Cat-PAD Treatment (2 Courses) (N=148) | Placebo (N=144)
Nasopharyngitis (Infections and infestations) | 15 (19) | 20 (30) | 18 (36)
Sinusitis (Infections and infestations) | 6 (6) | 6 (9) | 5 (7)
Influenza (Infections and infestations) | 5 (8) | 4 (4) | 7 (11)
Upper respiratory tract infection (Infections and infestations) | 2 (4) | 2 (2) | 8 (10)
Bronchitis (Infections and infestations) | 4 (4) | 4 (4) | 2 (2)
Tonsillitis (Infections and infestations) | 3 (3) | 3 (4) | 2 (2)
Pharyngitis (Infections and infestations) | 1 (1) | 4 (5) | 1 (1)
Conjunctivitis (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (2) | 5 (5)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 6 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 3 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (4) | 3 (5)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 5 (21) | 6 (6) | 6 (7)
Migraine (Nervous system disorders) | 1 (1) | 1 (2) | 6 (7)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
To avoid disclosures that may affect the proprietary rights of the Sponsor, the Investigator agrees to allow Circassia the opportunity to review all manuscripts and abstracts 60 days prior to submission for publication. Circassia reserves the right to include the report of this study in any regulatory documentation or submission or in any informational materials.

DOCUMENTS (2):
  • Study Protocol (2014-12-08): https://cdn.clinicaltrials.gov/large-docs/44/NCT02040844/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-23): https://cdn.clinicaltrials.gov/large-docs/44/NCT02040844/SAP_001.pdf